CLINICAL TRIAL: NCT05943561
Title: Biomarkers in Concussion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Nicholas Streicher, Principle Investigator, Medstar Health Research Institute
Other Study IDs: STUDY00006198
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Concussion, Mild; Concussion, Intermediate; Concussion, Severe
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concussion: Has an acute concussion
- Non-concussion: Does not have a concussion

SUMMARY:
This will be an observational study measuring serum Neurofilament Light Chain concentrations and associated symptoms, with a control branch, and a post-concussion branch.

ELIGIBILITY:
Inclusion Criteria:

Over 12 years of age Athletes participating on a sports team willing to participate; undergo blood draws either weekly or every two weeks, depending on arm of study.

Exclusion criteria:

Existing active neurodegenerative disorder (ie severe TBI) Active peripheral nerve disorder (ie diabetic neuropathy)

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Athletes with or without concussion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Normalization of NfL levels | 12 weeks

SECONDARY OUTCOMES:
Resolution of concussion symptoms | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Streicher, Principal Investigator — Medstar Health Research Institute

IPD SHARING:
Plan to Share IPD: No